CLINICAL TRIAL: NCT04508751
Title: Fetal Body Composition and Free-Breathing Magnetic Resonance Imaging
Brief Title: PED NEONAT 20-000599 Fetal Body Composition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Katie Strobel, MD, Principle Investigator, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-000599
Record Dates: First submitted 2020-08-03; First posted 2020-08-11 (Actual); Results first posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2022-10

CONDITIONS: IUGR; Gestational Diabetes; Pregnancy Related
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Pregnant mothers who's infants were diagnosed with intrauterine growth restriction and mothers with pregnancies complicated by gestational diabetes, and mothers with healthy uncomplicated pregnancies will be recruited to have a fetal MRI in the third trimester.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Pregnancy (Other): Patient will have a fetal MRI performed in the third trimester. All MRI scans will be performed on 3 T scanners (e.g., Skyra or Prisma, Siemens). Our newly developed FB-MRI quantification technique leverages a multi-echo 3D stack-of-radial sampling trajectory with golden-angle acquisition ordering to suppress motion artifacts and enable free-breathing imaging of the abdomen in around 5 minutes. In addition, our FB-MRI technique is compatible with data under sampling to accelerate the free-breathing scan to 1-2 min. In this study, we will optimize the parameters of our FB-MRI technique (spatial resolution, spatial coverage, acceleration factor) to balance trade-offs between scan time, image quality, fat quantification accuracy, and patient comfort/compliance. Subjects will be provided ear plugs to limit amount of noise from MRI machines.
  Maternal demographics, pregnancy clinical course and infant growth parameters will be recorded.
  Interventions: Other: 3T "Free-Breathing" Fetal Magnetic Resonance Imaging
- Pregnant Mothers with gestational diabetes (Other): Patient will have a fetal MRI performed in the third trimester. All MRI scans will be performed on 3 T scanners (e.g., Skyra or Prisma, Siemens). Our newly developed FB-MRI quantification technique leverages a multi-echo 3D stack-of-radial sampling trajectory with golden-angle acquisition ordering to suppress motion artifacts and enable free-breathing imaging of the abdomen in around 5 minutes. In addition, our FB-MRI technique is compatible with data under sampling to accelerate the free-breathing scan to 1-2 min. In this study, we will optimize the parameters of our FB-MRI technique (spatial resolution, spatial coverage, acceleration factor) to balance trade-offs between scan time, image quality, fat quantification accuracy, and patient comfort/compliance. Subjects will be provided ear plugs to limit amount of noise from MRI machines.
  Maternal demographics, pregnancy clinical course and infant growth parameters will be recorded.
  Interventions: Other: 3T "Free-Breathing" Fetal Magnetic Resonance Imaging
- Pregnant Mothers with infants diagnosed with IUGR (Other): Patient will have a fetal MRI performed in the third trimester. All MRI scans will be performed on 3 T scanners (e.g., Skyra or Prisma, Siemens). Our newly developed FB-MRI quantification technique leverages a multi-echo 3D stack-of-radial sampling trajectory with golden-angle acquisition ordering to suppress motion artifacts and enable free-breathing imaging of the abdomen in around 5 minutes. In addition, our FB-MRI technique is compatible with data under sampling to accelerate the free-breathing scan to 1-2 min. In this study, we will optimize the parameters of our FB-MRI technique (spatial resolution, spatial coverage, acceleration factor) to balance trade-offs between scan time, image quality, fat quantification accuracy, and patient comfort/compliance. Subjects will be provided ear plugs to limit amount of noise from MRI machines.
  Maternal demographics, pregnancy clinical course and infant growth parameters will be recorded.
  Interventions: Other: 3T "Free-Breathing" Fetal Magnetic Resonance Imaging

INTERVENTIONS:
Other: 3T "Free-Breathing" Fetal Magnetic Resonance Imaging — Subject will have a one time MRI scan.

SUMMARY:
Obesity is an ongoing public health problem that is difficult to treat. There is evidence that obesity has fetal origins. Body composition, including visceral, subcutaneous, brown, and hepatic fat have been found to be important predictors in obesity and metabolic syndrome. Magnetic resonance imaging (MRI) can quantify body composition that does not require radiation but is motion limited. The investigators have developed a motion-compensated MRI sequence, also known as "free breathing" MRI. In this study, the investigators plan to obtain free-breathing MRIs of pregnant women in the third trimester of pregnancy. MRIs will be obtained from healthy mothers, mothers with growth-restricted fetuses, and mothers with gestational diabetes. The different types of adipose tissue will be measured and compared between groups and correlated to birth growth parameters. The goal is this study is to assess if motion-compensated MRI can help predict early growth patterns in infancy.

DETAILED DESCRIPTION:
1.1 OBJECTIVE This study's goals are to: 1) use free-breathing magnetic resonance imaging (FB-MRI) to measure fetal body composition in the third trimester and 2) determine how the FB-MRI quantitative measurements compare to growth parameters at birth.

1.2 HYPOTHESES AND SPECIFIC AIMS

To accomplish the investigators' objectives, the aims and hypotheses are as follows:

Specific Aim 1:

In a prospective study in women with healthy pregnancies and women with fetuses that have intrauterine growth restriction (IUGR) and gestational diabetes, the investigators will quantify fetal subcutaneous, visceral, and brown adipose tissue volumes and proton-density fat fraction (PDFF) using FB-MRI in the third trimester.

Hypothesis 1: Using a FB-MRI technique the investigators will find the following,

1. The growth-restricted fetus will have less visceral, subcutaneous, and brown adipose tissue volume and PDFF when compared to healthy fetuses and fetuses whose mothers have gestational diabetes.
2. Fetuses whose mothers have gestational diabetes will have a greater subcutaneous and visceral adipose tissue volume and PDFF compared to healthy fetuses.

Specific Aim 2:

In a prospective study in pregnant women and their fetuses, the investigators will compare volume and PDFF measurements of fetal visceral, subcutaneous, and brown adipose tissue obtained with FB-MRI to birth growth parameters of these infants.

Hypothesis 2: The volume and PDFF of fetal visceral and subcutaneous adipose tissue will correlate positively with birth weight and length z-score.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with singleton pregnancies (healthy cohort)
* Pregnant women with fetuses with weights < 10th percentile weight for gestational age (IUGR cohort)
* Pregnant women with gestational diabetes (diabetes cohort)

Exclusion Criteria:

* Pregnant minors
* Major congenital anomalies or disease processes in the fetus
* Fetus with known chromosomal anomalies
* Mothers who do not plan to deliver at UCLA
* Multiple pregnancy (i.e. twins, triplets, etc)
* History of claustrophobia
* Contraindications to MRI such as metallic devices in the body that are not MRI compatible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified female patients who are pregnant
Enrollment: 23 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2022-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California-Los Angeles, Los Angeles, California
  - University of California- Los Angeles Santa Monica, Santa Monica, California

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited by study investigator or obstetrician through medical clinic.
Pre-assignment Details: One subject was excluded due to inability to schedule MRI scan
Groups:
- Healthy Pregnancy; Pregnant Mothers With Gestational Diabetes; Pregnant Mothers With Infants Diagnosed With IUGR: Patient will have a fetal MRI performed in the third trimester. All MRI scans will be performed on 3 T scanners (e.g., Skyra or Prisma, Siemens). Our newly developed FB-MRI quantification technique leverages a multi-echo 3D stack-of-radial sampling trajectory with golden-angle acquisition ordering to suppress motion artifacts and enable free-breathing imaging of the abdomen in around 5 minutes. In addition, our FB-MRI technique is compatible with data under sampling to accelerate the free-breathing scan to 1-2 min. In this study, we will optimize the parameters of our FB-MRI technique (spatial resolution, spatial coverage, acceleration factor) to balance trade-offs between scan time, image quality, fat quantification accuracy, and patient comfort/compliance. Subjects will be provided ear plugs to limit amount of noise from MRI machines.
  Maternal demographics, pregnancy clinical course and infant growth parameters will be recorded.
  3T "Free-Breathing" Fetal Magnetic Resonance Imaging: Subject will have a one time MRI scan.
Period: Overall Study
Arm/Group | Healthy Pregnancy | Pregnant Mothers With Gestational Diabetes | Pregnant Mothers With Infants Diagnosed With IUGR
Started | 10 | 5 | 7
Completed | 10 | 5 | 5
Not Completed | 0 | 0 | 2
Not completed — Discontinued study early due to maternal discomfort | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Healthy Pregnancy: Pregnancy without fetal anatomic or chromosomal abnormalities, FGR, or GDM.
- Pregnant Mothers With Gestational Diabetes: GDM was defined as a positive glucola screen at 26 to 32 weeks gestation.
- Pregnant Mothers With Infants Diagnosed With IUGR: IUGR was defined as fetal weight and abdominal circumference <10th percentile on ultrasound for a given gestational age or per obstetrician documentation on at least two medical notes
- Total: Total of all reporting groups
Arm/Group | Healthy Pregnancy | Pregnant Mothers With Gestational Diabetes | Pregnant Mothers With Infants Diagnosed With IUGR | Total
Number analyzed (Participants) | 10 | 5 | 5 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34.5 [29.8 to 38] | 33 [30.5 to 36.5] | 35 [27.5 to 36] | 34.5 [29.25 to 36.75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 5 | 20
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 1 | 7
  Not Hispanic or Latino | 8 | 1 | 4 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 5 | 3 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 5 | 20
Glucose tolerance test at 1 hour [Median (Inter-Quartile Range); unit: mg/dL] | 87 [62 to 112] | 182 [157 to 191] | 131 [102 to 146] | 109 [73 to 151]

OUTCOME MEASURES:

1. Primary Outcome: Maternal Visceral Adipose Tissue Volume
Description: MRI data will be reconstructed by Siemens scanner software to produce 3D fat-water separated images and PDFF maps. The FB-MRI radial data will be transferred to a separate workstation for custom reconstruction of 3D fat-water-separated images and PDFF maps and analysis. Visceral adipose tissue PDFF values will be directly measured from regions of interest.
Time Frame: During the procedure (MRI)
Measure: Median (Inter-Quartile Range); unit: mm3
Arm/Group | Healthy Pregnancy | Pregnant Mothers With Gestational Diabetes | Pregnant Mothers With Infants Diagnosed With IUGR
Number analyzed (Participants) | 10 | 5 | 5
mm3 | 97593 [78014 to 121081] | 169626 [137736 to 227035] | 96787 [82327 to 184784]

2. Primary Outcome: Fetal Liver PDFF
Description: MRI data will be reconstructed by Siemens scanner software to produce 3D fat-water separated images. The distribution/extent of hepatic fat will be manually delineated/drawn on the 3D MRI images and PDFF maps. This work will be performed by PI Strobel with validation from PI Wu.
Time Frame: During the procedure (MRI)
Measure: Median (Inter-Quartile Range); unit: percentage of triglycerides/
Arm/Group | Healthy Pregnancy | Pregnant Mothers With Gestational Diabetes | Pregnant Mothers With Infants Diagnosed With IUGR
Number analyzed (Participants) | 10 | 5 | 5
percentage of triglycerides/ | 3.2 [3.0 to 3.3] | 5.2 [4.2 to 5.5] | 1.9 [1.4 to 3.7]

3. Secondary Outcome: Fetal Subcutaneous Tissue Volume
Description: MRI data will be reconstructed by Siemens scanner software to produce 3D fat-water separated images and PDFF maps. The FB-MRI radial data will be transferred to a separate workstation for custom reconstruction of 3D fat-water-separated images and PDFF maps and analysis. Subcutaneous adipose tissue PDFF values will be directly measured from regions of interest.
Time Frame: During the procedure (MRI)
Measure: Median (Inter-Quartile Range); unit: mm3
Arm/Group | Healthy Pregnancy | Pregnant Mothers With Gestational Diabetes | Pregnant Mothers With Infants Diagnosed With IUGR
Number analyzed (Participants) | 10 | 5 | 5
mm3 | 241 [232 to 255] | 280 [261 to 295] | 220 [205 to 235]

4. Secondary Outcome: Maternal Subcutaneous Tissue Volume
Description: MRI data will be reconstructed by Siemens scanner software to produce 3D fat-water separated images. The distribution/extent of subcutaneous fat will be manually delineated/drawn on the 3D MRI images and PDFF maps and used to calculate volume of subcutaneous adipose tissue. This work will be performed by PI Strobel with validation from PI Wu.
Time Frame: During the procedure (MRI)
Measure: Median (Inter-Quartile Range); unit: mm3
Arm/Group | Healthy Pregnancy | Pregnant Mothers With Gestational Diabetes | Pregnant Mothers With Infants Diagnosed With IUGR
Number analyzed (Participants) | 10 | 5 | 5
mm3 | 157319 [126300 to 200028] | 216264 [161461 to 325975] | 159197 [84024 to 339707]

5. Secondary Outcome: Maternal Hepatic Fat PDFF
Description: MRI data will be reconstructed by Siemens scanner software to produce 3D fat-water separated images and PDFF maps. The FB-MRI radial data will be transferred to a separate workstation for custom reconstruction of 3D fat-water-separated images and PDFF maps and analysis. Hepatic adipose tissue PDFF values will be directly measured from regions of interest.
Time Frame: During the procedure (MRI)
Measure: Median (Inter-Quartile Range); unit: % triglycerides
Arm/Group | Healthy Pregnancy | Pregnant Mothers With Gestational Diabetes | Pregnant Mothers With Infants Diagnosed With IUGR
Number analyzed (Participants) | 10 | 5 | 5
% triglycerides | 2.1 [1.8 to 2.8] | 3.2 [2.1 to 3.8] | 2.2 [1.1 to 5.0]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Healthy Pregnancy | Pregnant Mothers With Gestational Diabetes | Pregnant Mothers With Infants Diagnosed With IUGR
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/10 | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Because this is a pilot study, our sample size is limited, and the results should be considered exploratory. We did not longitudinally measure body composition during pregnancy and infancy. Future follow-up would be required to understand if maternal and fetal body composition are truly associated with future childhood and adulthood obesity and various metabolic complications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT04508751/Prot_SAP_000.pdf